CLINICAL TRIAL: NCT00611000
Title: Effect of Folate on Colonic and Blood Cells
Brief Title: Effect of Folate on DNA in Colon Tissue and Blood Samples From Patients at Increased Risk of Developing Colorectal Neoplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: Single | Purpose: Prevention
Other Study IDs: CDR0000582113; RUH-PHO-0514-0306
Record Dates: First submitted 2008-02-07; First posted 2008-02-08 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folic Acid; DNA Methylation; Gene Expression Profiling; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Dietary Supplement: folic acid
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients at risk of cancer in the laboratory may help doctors learn more about the effect of folate on DNA and identify biomarkers related to cancer.

PURPOSE: This phase I trial is studying the effect of folate on DNA in colon tissue and peripheral blood samples from patients at increased risk of developing colorectal neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To analyze the effects of changes in levels of dietary folate intake on damage to DNA and repair capacity, mRNA expression, and DNA uracil incorporation in peripheral blood mononuclear cell and rectal biopsy cell samples from patients at increased risk for developing colorectal neoplasia.

OUTLINE: Patients are enrolled into 1 of 2 intervention groups..

* Group I (folate depletion [in-patient]): Patients consume a weight-maintaining, average folate diet with no high folate-containing foods for 8 weeks. Patients are then admitted to The Rockefeller University Hospital and placed on a weight-maintaining, low-folate diet for 12 weeks. During the last 4 weeks of the in-patient period, patients receive oral folic acid supplementation once daily for 4 weeks.
* Group II (folate supplementation [out-patient]): Patients consume a weight-maintaining, average folate diet with no high folate-containing foods for 16 weeks as an out-patient. After the first 8 weeks of the diet, patients also receive oral folic acid supplementation once daily for 8 weeks.

Patients undergo blood sample collection periodically for biomarker correlative studies. Samples are analyzed for serum and red cell folate and homocystine levels to assess folate depletion; methylentetrahydrofolate reductase (MTHFR) polymorphism to test for inherited alterations of folate metabolism; serum and plasma biomarkers; and DNA studies. Patients also undergo tissue sample collection by sigmoidoscopy and rectal biopsy periodically. Tissue samples are assessed for mucosal folate concentration and mucosal folic acid metabolites; DNA methylation; and gene assays by microarray analysis.

After completion of study intervention, patients are followed at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk for developing colorectal neoplasia due to 1 of the following:

  * Personal history of colorectal adenomatous polyps
  * Family history of colorectal adenoma or adenocarcinoma
* No hereditary nonpolyposis colorectal cancer (HNPCC)
* No more than one first-degree family member with colorectal or endometrial malignancies

PATIENT CHARACTERISTICS:

* Ambulatory
* Female patients must be ≥ 2 years post-menopausal (i.e., 2 years after the last menstrual period)
* Negative pregnancy test
* Male patients must use effective contraception during and for 2 months after completion of study treatment (for male patients enrolled in the folate depletion group)
* Serum folate level ≤ 20 ng/mL
* Plasma vitamin B12 level ≥ 250 pg/mL
* Serum homocysteine level ≤ 17 μmol/L
* ALT or AST ≤ 2 times upper limit of normal
* No unexplained elevated alkaline phosphatase
* Creatinine ≤ 2.0 mg/dL
* HIV negative
* No folate metabolism abnormalities or predisposing conditions
* No prior malignancy except nonmelanoma skin cancer
* No intestinal malabsorption or inflammatory bowel disease
* No excessive bleeding or coagulation disorder
* No untreated hyperthyroidism
* No diabetes mellitus requiring insulin
* No daily alcohol intake > 2 ½ shot glasses of whisky or three 8-ounce glasses of beer or wine
* No sustained blood pressure > 150/95 mm Hg for three consecutive readings
* No other serious illness that would limit life expectancy to < 6 months

PRIOR CONCURRENT THERAPY:

* No prior gastrointestinal surgery, including gastrectomy or small or large bowel resections

  * Prior appendectomy or surgery of the esophagus allowed
* More than 3 months since regular ingestion of ≥ 650 mg of aspirin (≥ 2 tablets of 325 mg regular strength OR > 1 tablet of 500 mg extra strength aspirin) per day

  * The following drugs are allowed for cardiovascular prophylaxis provided the patient has been taking the drug regularly for ≥ 1 month and continues to take the same dose during study participation:

    * One or two regular strength aspirin tablets (i.e., 325 mg per tablet) per day
    * One baby aspirin tablet (81 mg tablet) per day
* More than 3 months since regular daily ingestion of other non-steroidal anti-inflammatory drugs (NSAIDs)
* No concurrent anticoagulation therapy
* No concurrent sterol-binding resins, such as cholestyramine (for the treatment of high blood cholesterol)
* No other concurrent investigational drugs
* No other concurrent medications that might, in the view of the study physicians, alter rectal mucosal proliferation, folate metabolism, or renal/hepatic metabolism
* No concurrent weight control medications
* No concurrent supplemental folate preparation containing > 400 mcg of folic acid per day
* No concurrent hormone replacement therapy, including oral, transplanted, or injected contraceptives

  * Concurrent thyroid hormone replacement allowed provided the patient is euthyroid
* No concurrent medication interfering with folic acid metabolic effects, including any of the following:

  * Methotrexate
  * Phenytoin
  * Phenobarbital
  * Primidone
  * Sulfonamides
  * Folinic acid derivatives
* No concurrent lipid-lowering medications other than usual doses of the class of drugs known as statins

  * The following statin drugs are allowed provided the patient has been taking the drug regularly for ≥ 1 month and continues to take the same dose during study participation:

    * Atorvastatin (10 or 20 mg/day)
    * Fluvastatin (20 mg or 40 mg/day)
    * Lovastatin (10 or 20 mg/day)
    * Pravastatin (10 or 20 mg/day)
    * Simvastatin (5 or 10 mg/day)

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-06; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
DNA uracil incorporation in peripheral blood mononuclear cells (PBMCs)
Strand breaks in the coding region of p53 in PBMCs and rectal biopsy cells
DNA methylation (overall, p53 coding, p16 promoter, MLH1 promoter) in PBMCs and rectal biopsy cells

SECONDARY OUTCOMES:
Differential gene expression in colonic and PBMCs by microarray analysis

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Holt, MD, Principal Investigator — Rockefeller University